CLINICAL TRIAL: NCT00974142
Title: A Randomized, Double-Blinded, Placebo-Controlled Protocol of Oral Cyclosporine in Patients With Advanced Stage Chronic Obstructive Pulmonary Disease
Brief Title: Oral Cyclosporine in Chronic Obstructive Pulmonary Disease
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Michael Donahoe (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor-Investigator, Michael Donahoe, Professor, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PRO09050330
Record Dates: First submitted 2009-09-09; First posted 2009-09-10 (Estimated); Results first posted 2018-05-09 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2018-04

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: COPD; Chronic Obstructive Pulmonary Disease; Cyclosporine; Oral Immunotherapy; Advanced stage
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Cyclosporine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cyclosporine (Experimental)
  Interventions: Drug: Cyclosporine
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Cyclosporine — Fifteen patients will receive cyclosporine at an initial dosing of 3.0 mg/kg/day.
  Other Names: Neoral
  Arms: Cyclosporine
Drug: Placebo — Fifteen patients will receive will receive placebo.
  Arms: Placebo

SUMMARY:
This is a randomized, double-blinded, placebo-controlled trial of oral Cyclosporine A (CsA) in patients with advanced stage chronic obstructive pulmonary disease. The purpose of the study is to evaluate the safety and effectiveness of CsA as a therapy for the adaptive immune response in advanced stage Chronic Obstructive Pulmonary Disease (COPD).

Subjects between 45 and 80 years of age with a confirmed diagnosis of advanced stage COPD, not responsive to conventional inhaler therapy, who meet all the study requirements, will be enrolled in this study. A total of 30 subjects of either sex will be enrolled in this study.

ELIGIBILITY:
Inclusion Criteria:

* Age between 45 and 80 years
* A confirmed diagnosis of advanced stage COPD, using current accepted diagnostic criteria, including clinical/laboratory findings, pulmonary function tests, and appropriate history to exclude other disorders that could explain their lung disease. The accepted range of forced expiratory volume at one second will include 25% ≤ forced expiratory volume at one second ≤ 60%
* Subjects agree to maintain a stable medication regimen in the absence of a disease flare
* Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1, or 2
* carbon dioxide partial pressure < 45 mm Hg, room air oxyhemoglobin saturation > 85%
* A willingness to participate in all portions of the protocol, including serial bronchoscopy, requisite surveillances, and ancillary immunologic studies in follow-up visits at this institution
* For woman of childbearing age, a negative pregnancy test, and a willingness to use two methods of contraception, or abstinence
* An ability and willingness to provide written informed consent

Exclusion Criteria:

* Three, or more exacerbations of lower respiratory disease in the past year requiring systemic corticosteroids, or one exacerbation requiring hospitalization in the past 6 months
* Intubation for COPD, or other cause of respiratory failure in the past year
* Use of immunosuppressive therapy including oral prednisone > 10mg per day other than aerosolized corticosteroids, anytime within three months prior to participation
* Evidence for an opportunistic infection/colonization of the airways, i.e., non-bacterial
* Evidence for systemic illness including hematologic disorders (defined by an absolute neutrophil count (ANC) < 4000 /mL and platelets < 120,000/mL), cirrhosis, or hepatic insufficiency (total bilirubin, or alkaline phosphatase > 1.5 x normal, serum glutamate oxaloacetate transaminase, or serum glutamate pyruvate transaminase > 1.2 x normal values), or a coagulopathy (INR > 1.4), seizure disorder
* Evidence for renal insufficiency with a calculated creatinine clearance using the Cockcroft and Gault's method of < 80 ml/min for males and < 70 ml/min for females, or serum creatinine > 1.4 mg/dL.
* Evidence of coronary artery disease by history, e.g., angina or history of myocardial infarction within the past 12 months, unless corrected by coronary artery bypass graft within < 5 years, and asymptomatic since
* Evidence for systemic abnormal renal function manifested by uncontrolled hypertension (systolic blood pressure > 160 mmHg or diastolic blood pressure >90 mmHg), hyperkalemia (serum potassium > 5.0 meq/dl, and/or elevated serum potassium above the normal range for the subject's age)
* Pregnancy or lactation, or inability to take contraception during and for 6 months following treatment
* Positive HIV, or hepatitis B or C serology, or another active infection
* Current or past history of cancer excluding basal or squamous cell skin cancer
* Undiagnosed pulmonary nodule requiring diagnostic evaluation
* Weight loss > 10% usual body weight over the past 6 months or a BMI < 18
* Known hypersensitivity or allergy to cyclosporine
* Concurrent participation in other clinical trials within the prior month
* Known medical or psychological condition (severe personality disorder or mental illness) that would not permit the subject to complete the trial or sign informed consent
* Autoimmune disorders or other disorders with suspected systemic immune involvement
* Active smoking history or urinary cotinine > 2
* Hypersensitivity to midazolam or narcotics which would not allow bronchoscopy sedation
* Concurrent use of drugs with a known interaction with cyclosporine

Ages: 45 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2009-09; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Donahoe, MD, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh, Pittsburgh, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited from local clinics, advertisement, and a disease specific registry
Pre-assignment Details: 772 patients underwent initial screening and 43 were eligible to sign consent. These patients underwent a second 2 week screening process and 17 subjects met all criteria for randomization
Groups:
- Cyclosporine: Randomized post 2nd level screen to 3 mg/kg / day oral cyclosporine
- Placebo: Randomized to placebo capsules identical in appearance to cyclosporine
Period: Overall Study
Arm/Group | Cyclosporine | Placebo
Started | 8 | 9
Completed | 8 | 9
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cyclosporine | Placebo | Total
Number analyzed (Participants) | 8 | 9 | 17
Age, Continuous [Median (Full Range); unit: years] | 68 [55 to 79] | 63 [48 to 77] | 67 [48 to 79]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 4 | 6
  Male | 6 | 5 | 11
Forced Vital Capacity (%) [Median (Inter-Quartile Range); unit: % predicted] | 88 [71 to 105] | 77 [60 to 94] | 79 [60 to 105]
Forced Expiratory Volume 1 second (%) [Median (Full Range); unit: % predicted] | 38 [31 to 54] | 43 [27 to 58] | 39 [27 to 58]
Functional Residual Capacity (%) [Median (Full Range); unit: % predicted] | 146 [108 to 180] | 149 [81 to 170] | 149 [81 to 180]
Total Lung Capacity (%) [Median (Full Range); unit: % predicted] | 123 [100 to 145] | 119 [84 to 138] | 119 [84 to 145]
Partial pressure of carbon dioxide (pCO2) [Mean (Standard Deviation); unit: mm Hg] | 40 (3.6) | 42.6 (3.9) | 41.2 (3.7)
Partial pressure of oxygen (pO2) [Mean (Standard Deviation); unit: mm Hg] | 71 (11) | 76 (20) | 74 (15)
Weight [Median (Full Range); unit: kilograms] | 83 [60 to 105] | 93 [55 to 119] | 84 [55 to 119]
Systolic blood pressure (mm Hg) [Median (Full Range); unit: mm Hg] | 141 [125 to 152] | 133 [104 to 150] | 138 [104 to 152]
Diastolic blood pressure (mm Hg) [Median (Full Range); unit: mm Hg] | 82 [71 to 95] | 78 [70 to 91] | 79 [70 to 95]
White blood cell count [Mean (Standard Deviation); unit: x10E ^09/L] | 7.3 (1.3) | 6.6 (2.0) | 7.1 (2.2)
Hemoglobin [Mean (Standard Deviation); unit: grams / dL] | 13.7 (1.0) | 13.6 (0.9) | 13.7 (1.03)
Blood Urea Nitrogen [Mean (Standard Deviation); unit: mg / dL] | 16 (5.4) | 13 (3.2) | 13.4 (3.9)
Creatinine [Mean (Standard Deviation); unit: mg / dL] | 0.9 (0.2) | 0.9 (0.2) | 0.9 (0.2)
Glucose [Mean (Standard Deviation); unit: mg / dL] | 102 (13) | 113 (29) | 111 (29)
Cholesterol [Mean (Standard Deviation); unit: mg / dL] | 183 (30) | 193 (20) | 183 (20)

OUTCOME MEASURES:

1. Primary Outcome: Safety Profile of Oral Cyclosporin A Immunotherapy in Advanced Stage Chronic Obstructive Pulmonary Disease Patients- Nephrotoxicity - Measured by Serum Creatinine
Description: Measurement of nephrotoxicity by monitoring serum creatinine over 16 week treatment interval. Mean serum creatinine values were assessed at Week 2, 4, 6, 8, 10, 12 and 16. The mean values of all measurements for each participant were calculated and then the mean across participants was calculated. Values expressed as mean ± SD.
Time Frame: 16 weeks
Measure: Mean (Standard Deviation); unit: mg / dL
Arm/Group | Cyclosporine | Placebo
Number analyzed (Participants) | 8 | 9
mg / dL | 0.94 (0.2) | 0.88 (0.2)

2. Primary Outcome: Safety Profile of Oral Cyclosporin A Immunotherapy in Advanced Stage Chronic Obstructive Pulmonary Disease Patients - Number of Patients That Developed Renal Insufficiency
Description: Development of renal insufficiency defined as > 30% elevation in serum creatinine above baseline which required dose modification of the cyclosporine over 16 week treatment interval at Week 2, 4, 6, 8, 10, 12 and 16. Outcome measured the number of subjects who developed renal insufficiency during the study treatment interval.
Time Frame: 16 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Cyclosporine | Placebo
Number analyzed (Participants) | 8 | 9
Participants | 4 | 1

3. Primary Outcome: Safety Profile of Oral Cyclosporin A Immunotherapy in Advanced Stage Chronic Obstructive Pulmonary Disease Patients - Number of Patients That Developed Infection Requiring Systemic Antibiotic Therapy
Description: Clinical diagnosis of infection which requires systemic antibiotic therapy during the 16 week study interval at Week 2, 4, 6, 8, 10, 12 and 16. Outcome measured the number of subjects who developed an infection requiring systemic antibiotic therapy during the study treatment interval.
Time Frame: 16 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Cyclosporine | Placebo
Number analyzed (Participants) | 8 | 9
Participants | 1 | 1

4. Secondary Outcome: Pharmacokinetic - Pharmacodynamic Relationship of Oral Cyclosporine and Biomarkers of an Adaptive Immune Response - Cyclosporine Blood Levels
Description: Cyclosporine blood levels on therapy over 16 week treatment interval were measured at Weeks 2, 4, 6, 8, 10, 12 & 16. The median for each participant was found and then the overall median was determined. Values expressed as median (full range).
Time Frame: 16 weeks
Population: Cyclosporine blood levels were not analyzed in placebo group.
Measure: Median (Full Range); unit: ng/mL
Arm/Group | Cyclosporine | Placebo
Number analyzed (Participants) | 8 | 0
ng/mL | 147 [69 to 196] |

5. Secondary Outcome: Peripheral Blood T Cell Biomarkers Over 16 Week Treatment Interval - Change in the Percentage of Cluster of Differentiation 4 (CD4)
Description: Outcome measured the change in the percentage of cluster of differentiation 4 (CD4) at midpoint assessment (Week 8) and at the conclusion of treatment (Week 16). Values expressed as median (full range).
Time Frame: at Week 8 and Week 16
Measure: Median (Full Range); unit: % of cells expressing biomarkers
Arm/Group | Cyclosporine | Placebo
Number analyzed (Participants) | 8 | 9
% of cells expressing biomarkers | -3.1 [-18.8 to 3.5] | 3.6 [-8.5 to 45.2]

6. Secondary Outcome: Peripheral Blood T Cell Biomarkers Over 16 Week Treatment Interval - Change in the Percentage of Cluster of Differentiation 8 and Cluster of Differentiation 28
Description: Outcome measured the change in the percentage of peripheral blood T cell biomarkers - cluster of differentiation 8 (CD8), cluster of differentiation 28 (CD28) at midpoint assessment (Week 8) and at the conclusion of treatment (Week 16). Values expressed as median (full range).
Time Frame: at Week 8 and Week 16
Measure: Median (Full Range); unit: % of cells expressing biomarkers
Arm/Group | Cyclosporine | Placebo
Number analyzed (Participants) | 8 | 9
% of cells expressing biomarkers | -0.78 [-19.2 to 6.3] | -1.6 [-6.6 to 3.0]

7. Secondary Outcome: Peripheral Blood T Cell Biomarkers Over Treatment Interval - Change in the Percentage of Cluster of Differentiation 8 and Major Histocompatibility Complex II
Description: Outcome measured the change in the percentage of peripheral blood cells expressing biomarker - cluster of differentiation 8 (CD8), major histocompatibility complex (MHC) II at midpoint assessment (Week 8) and at the conclusion of treatment (Week 16). Values expressed as median (full range).
Time Frame: at Week 8 and Week 16
Measure: Median (Full Range); unit: % of cells expressing biomarkers
Arm/Group | Cyclosporine | Placebo
Number analyzed (Participants) | 8 | 9
% of cells expressing biomarkers | -2.4 [-11.2 to 7.2] | 0.5 [-4.7 to 3.1]

8. Secondary Outcome: Peripheral Blood T Cell Biomarkers Over Treatment Interval - Change in the Percentage of Cluster of Differentiation 8+ Interferon Gamma
Description: Outcome measured the change in the percentage of peripheral blood T cell biomarkers - CD8+interferon gamma at midpoint assessment (Week 8) and at the conclusion of treatment (Week 16). Values expressed as median (full range).
Time Frame: at Week 8 and Week 16
Measure: Median (Full Range); unit: % of cells expressing biomarkers
Arm/Group | Cyclosporine | Placebo
Number analyzed (Participants) | 8 | 9
% of cells expressing biomarkers | -4.1 [-24.1 to 49.6] | 4.4 [-44.6 to 51.3]

9. Secondary Outcome: Peripheral Blood T Cell Biomarkers Over Treatment Interval - Change in the Percentage of Cluster of Differentiation 4+ Interleukin-2
Description: Outcome measured the change in the percentage of peripheral blood T cell biomarkers - cluster of differentiation 4+ interleukin-2 at midpoint assessment (Week 8) and at the conclusion of treatment (Week 16). Values expressed as median (full range).
Time Frame: at Week 8 and Week 16
Measure: Median (Full Range); unit: % of cells expressing biomarkers
Arm/Group | Cyclosporine | Placebo
Number analyzed (Participants) | 8 | 9
% of cells expressing biomarkers | -1.7 [-13.3 to 16.8] | 4.7 [-15.6 to 11.1]

10. Secondary Outcome: Peripheral Blood T Cell Biomarkers Over Treatment Interval - Change in the Percentage of Cluster of Differentiation 8+ Tumor Necrosis Factor
Description: Outcome measured the change in the percentage of peripheral blood T cell biomarkers - CD8+ tumor necrosis factor at midpoint assessment (Week 8) and at the conclusion of treatment (Week 16). Values expressed as median (full range).
Time Frame: at Week 8 and Week 16
Measure: Median (Full Range); unit: % of cells expressing biomarkers
Arm/Group | Cyclosporine | Placebo
Number analyzed (Participants) | 8 | 9
% of cells expressing biomarkers | 0.0 [-52.6 to 9.8] | 2.3 [-18 to 32.3]

11. Secondary Outcome: Effects of Cyclosporin A on Respiratory Function - Change in the Percentage of Post Predicted Value of Forced Vital Capacity
Description: Outcome measured the change in the percentage of post predicted value of forced vital capacity at midpoint assessment (Week 8) and at the conclusion of treatment (Week 16). Values expressed as median (full range).
Time Frame: at Week 8 and Week 16
Measure: Median (Full Range); unit: Percentage of post predicted value
Arm/Group | Cyclosporine | Placebo
Number analyzed (Participants) | 8 | 9
Percentage of post predicted value | -0.01 [-.04 to 0.6] | 0.07 [-0.3 to 0.2]

12. Secondary Outcome: Effects of Cyclosporin A on Respiratory Function - Change in the Percentage of Post Predicted Value of Forced Expiratory Volume in 1 Second
Description: Outcome measured the change in the percentage of post predicted value of forced expiratory volume in 1 second at midpoint assessment (Week 8) and at the conclusion of treatment (Week 16). Values expressed as median (full range).
Time Frame: at Week 8 and Week 16
Measure: Median (Full Range); unit: Percentage of post predicted value
Arm/Group | Cyclosporine | Placebo
Number analyzed (Participants) | 8 | 9
Percentage of post predicted value | -0.02 [-0.3 to 0.3] | -0.02 [-0.2 to 0.1]

13. Secondary Outcome: Effects of Cyclosporin A on Respiratory Function - Change in Exercise Capacity by a Shuttle Walk Distance Measured in Feet
Description: Measurement of exercise capacity by a shuttle walk distance measured in feet at midpoint assessment (Week 8) and at the conclusion of treatment (Week 16). The purpose of the shuttle walk test is to see how far and fast a patient can walk (without stopping for a rest) by following a series of time signals.Values expressed as median (full range).
Time Frame: at Week 8 and Week 16
Measure: Median (Full Range); unit: feet
Arm/Group | Cyclosporine | Placebo
Number analyzed (Participants) | 8 | 9
feet | 230 [170 to 450] | 220 [140 to 350]

14. Secondary Outcome: Effects of Cyclosporin A on Symptoms - Change in Scores on a Shortness of Breath Scale
Description: Scores on a shortness of breath scale (University of California at San Diego Dyspnea scale): shortness of breath questionnaire scores are summed as a total score ranging from 0-120 with higher scores indicating more severe breathlessness. Assessments were performed at midpoint assessment (Week 8) and at the conclusion of treatment (Week 16). Values expressed as median (full range).
Time Frame: at Week 8 and Week 16
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Cyclosporine | Placebo
Number analyzed (Participants) | 8 | 9
units on a scale | 39 [10 to 81] | 39 [4 to 85]

ADVERSE EVENTS:
Time Frame: Patients received the intervention over 16 weeks but were monitored for a total of 40 weeks
Arm/Group | Cyclosporine | Placebo
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/9
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/9
Other Adverse Events (participants affected / at risk) | 6/8 | 5/9
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cyclosporine (N=8) | Placebo (N=9)
Renal insufficiency (Renal and urinary disorders) | 4 (4) | 1 (1)
Gastrointestinal upset (Gastrointestinal disorders) | 4 (4) | 0 (0)
Hyperkalemia (Renal and urinary disorders) | 2 (2) | 0 (0)
Hypertension (Renal and urinary disorders) | 1 (1) | 0 (0)
Tremor (Nervous system disorders) | 1 (1) | 0 (0)
Muscle cramp (Nervous system disorders) | 1 (1) | 0 (0)
Respiratory colonization (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) — Development of new respiratory system colonization without evidence for infection
Respiratory Infection -Bronchitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pulmonary nodule (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No